CLINICAL TRIAL: NCT04656028
Title: Impact of Genetic Testing and Motivational Counseling on the Adherence to Healthy Lifestyle and Hypolipidemic Therapy and Efficiency of Cascade Screening in Patients With Familial Hypercholesterolemia (GENMOTIV-FH)
Brief Title: Genetic Testing and Motivational Counseling for FH
Acronym: GENMOTIV-FH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-03/19
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hypercholesterolemia, Familial; Hypercholesterolemia, Familial, 1; Hypercholesterolemia, Familial, 2; Hypercholesterolemia, Familial, 3; Hypercholesterolemia, Familial, 4; Hypercholesterolemia, Familial, 4, Autosomal Recessive; Familial Hypercholesterolemia With Hyperlipemia; Hypercholesterolemia, Autosomal Dominant, Type B; Hypercholesterolemia, Autosomal Dominant; Hypercholesterolemia, Autosomal Dominant, 3; Apolipoprotein B-100, Familial Defective; Genetic Testing; Motivational Interviewing; Therapeutic Adherence; Therapeutic Adherence and Compliance; Treatment Adherence; Medication Adherence; Treatment Adherence and Compliance; Patient Adherence; Compliance; Patient Compliance; Familial Hypercholesterolemia; Familial Hypercholesterolemia - Heterozygous; Adherence, Patient; Adherence, Medication; Adherence
Keywords: Familial Hypercholesterolemia; FH; genetic testing; motivational counseling; motivational interviewing; cascade screening; adherence; compliance; Hypercholesterolemia, Familial; Hypercholesterolemia, Familial, 1; Hypercholesterolemia, Familial, 2; Hypercholesterolemia, Familial, 3; Hypercholesterolemia, Familial, 4; Hypercholesterolemia, Familial, 4, Autosomal Recessive; Familial Hypercholesterolemia with Hyperlipemia; Hypercholesterolemia, Autosomal Dominant, Type B; Hypercholesterolemia, Autosomal Dominant; Hypercholesterolemia, Autosomal Dominant, 3; Apolipoprotein B-100, Familial Defective; Therapeutic Adherence; Therapeutic Adherence and Compliance; Patient Adherence; Familial Hypercholesterolemia - Heterozygous; psychological counseling; Adherence, Patient; Adherence, Medication; Treatment Adherence; Medication Adherence; Treatment Adherence and Compliance; Patient Compliance
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia, Autosomal Dominant, 3; Hyperlipoproteinemia Type III; Hypercholesterolemia; Treatment Adherence and Compliance; Medication Adherence; Patient Compliance | interventions — Genetic Testing; Motivational Interviewing; Referral and Consultation; Diet

STUDY DESIGN:
Intervention Model Description: The trial is a randomized prospective cohort study. The study will include patients 18 years of age and older with a probable or definite diagnosis of FH according to the Dutch criteria (6 points or more). A total of 180 patients will be included in the study. All patients will be randomly divided into 2 groups for genetic testing. Randomization will be performed as block randomization with a 2:1 allocation ratio (2 with genetic testing : 1 without genetic testing). The allocation ratio 2:1 was chosen because in the group with genetic testing there will be cases where mutation(s) associated with FH will be identified and cases where the mutation(s) will not be identified. A separate analysis is planned in patients with genetic testing and identified mutation(s) and in patients with genetic testing but no identified mutation(s).
  Each study group will be randomized into 2 subgroups depending on the conduct of motivational counseling with an 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 - without genetic testing; subgroup without motivational counseling (Active Comparator): Group 1 - without genetic testing; subgroup without motivational counseling
  Interventions: Diagnostic Test: Lipid analysis; Other: Consultation with a cardiologist-lipidologist (correction of therapy, lifestyle, diet); Other: Visit 1; Other: Visit 2; Other: Visit 3; Other: Visit 4
- Group 1 - without genetic testing; subgroup with motivational counseling (Experimental): Group 1 - without genetic testing; subgroup with motivational counseling
  Interventions: Behavioral: Motivational Counseling; Diagnostic Test: Lipid analysis; Other: Consultation with a cardiologist-lipidologist (correction of therapy, lifestyle, diet); Other: Visit 1; Other: Visit 2; Other: Visit 3; Other: Visit 4
- Group 2 - with genetic testing; subgroup without motivational counseling (Experimental): Group 2 - genetic testing has been performed; subgroup without motivational counseling.
  Interventions: Genetic: Genetic Testing; Diagnostic Test: Lipid analysis; Other: Consultation with a cardiologist-lipidologist (correction of therapy, lifestyle, diet); Other: Visit 1; Other: Visit 2; Other: Visit 3; Other: Visit 4
- Group 2 - with genetic testing; subgroup with motivational counseling (Experimental): Group 2 - genetic testing has been performed; subgroup with motivational counseling.
  Interventions: Genetic: Genetic Testing; Behavioral: Motivational Counseling; Diagnostic Test: Lipid analysis; Other: Consultation with a cardiologist-lipidologist (correction of therapy, lifestyle, diet); Other: Visit 1; Other: Visit 2; Other: Visit 3; Other: Visit 4

INTERVENTIONS:
Genetic: Genetic Testing — DNA is extracted using the QIAamp® DNA Blood Mini Kit (Qiagen, Germany). The DNA concentration is measured on a Qubit 4.0 fluorometer (Thermo Fisher Scientific, USA (TFS)). NGS is performed on Nextseq 550 (Illumina, San Diego, CA, USA). The library preparation is performed using the SeqCap EZ Prime Choice Library kit (Roche, Basel, Switzerland). The Roche panel is used, consisting of 244 (CDS + 25 bp padding) genes including LDLR, APOB, and PCSK9. Reads are aligned to the reference genome (GRCh37). Sequencing analysis resultes in fastq files. Data processing is performed with BWA, Picard, bcftools, GATK3 and generally followed the GATK best practices for variant calling. For clinical interpretation, genetic variants with frequencies in the gnomAD database <0.5% are selected. The pathogenicity of variants is assessed according to the ACMG / AMP2015 guidelines. The identified SNPs are validated by Sanger sequencing (3500 DNA Analyzer, TFS).
  Arms: Group 2 - with genetic testing; subgroup with motivational counseling; Group 2 - with genetic testing; subgroup without motivational counseling
Behavioral: Motivational Counseling — Motivational counseling will be carried out during Visit 2 and in one month after Visit 2 by certified psychologist with taking into account the results of the psychodiagnostic survey conducted at the first and second visits.
  The goals of motivational counseling:
  1. Increasing motivation for a healthy lifestyle;
  2. Increasing adherence to treatment;
  3. Increased motivation to invite relatives for cascade screening. Motivational counseling will be carried out using methods of motivational interviewing, transtheoretical model of changes, cognitive-behavioral therapy, extended preventive counseling.
  Other Names: Motivational Interviewing
  Arms: Group 1 - without genetic testing; subgroup with motivational counseling; Group 2 - with genetic testing; subgroup with motivational counseling
Diagnostic Test: Lipid analysis — Assessment of total cholesterol, low density lipoproteins, high density lipoproteins, triglycerides, alanine aminotransferase.
Other: Consultation with a cardiologist-lipidologist (correction of therapy, lifestyle, diet) — All patients will be prescribed ezetimibe and statins (atorvastatin / rosuvastatin) at the maximum dosage. If somebody has an intolerance to atorvastatin, the drug will be replaced with rosuvastatin and vice versa. In case of intolerance to all drugs from the statin group, the patient will be prescribed ezetimibe with a PCSK9 inhibitor (alirocumab / evolocumab). After receiving the results of the lipid spectrum, ALT, if necessary, the lipid-lowering therapy may be corrected.
Other: Visit 1 — Visit 1: initially (on enrollment) - informed consents signing; lipid blood tests, patient data gathering, and consultation of cardiologist-lipidologist for optimization of lipid-lowering therapy and lifestyle; filling all questionnaires. After this visit patients are randomized to groups with or without genetic testing and then randomized to groups with or without motivational counseling.
  Each visit consists of two patient's attendances to the medical center. At the first attendance, it is planned to take blood for analysis, fill out questionnaires; at the second attendance - to perform, a consultation with a cardiologist-lipidologist according to the results of blood analysis. The time interval between two attendances is ≤ 7 days.
Other: Visit 2 — Visit 2 (in 2-3 months): lipid blood tests, patient data gathering, and consultation of cardiologist-lipidologist for optimization of lipid lowering-therapy and lifestyle; filling all questionnaires. Patients from the group with genetic testing will get the result of this genetic testing. Patients from the group with motivational counseling will get two consultations with a psychologist (motivational counseling on lifestyle modification) during Visit 2 and in one month after Visit 2.
  Each visit consists of two patient's attendances to the medical center. At the first attendance, it is planned to take blood for analysis, fill out questionnaires; at the second attendance - to perform a consultation with a cardiologist-lipidologist according to the results of blood analysis. The time interval between two attendances is ≤ 7 days
Other: Visit 3 — Visit 3 (in 3 months after Visit 2): lipid blood tests, patient data gathering, and consultation of cardiologist-lipidologist for optimization of lipid-lowering therapy and lifestyle; filling all questionnaires.
  Each visit consists of two patient's attendances to the medical center. At the first attendance, it is planned to take blood for analysis, fill out questionnaires; at the second attendance - to perform a consultation with a cardiologist-lipidologist according to the results of blood analysis. The time interval between two attendances is ≤ 7 days.
Other: Visit 4 — Visit 4 (in 12 months after Visit 3): lipid blood tests, patient data gathering, and consultation of cardiologist-lipidologist for optimization of lipid-lowering therapy and lifestyle; filling all questionnaires.
  Each visit consists of two patient's attendances to the medical center. At the first attendance, it is planned to take blood for analysis, fill out questionnaires; at the second attendance - to perform a consultation with a cardiologist-lipidologist according to the results of blood analysis. The time interval between two attendances is ≤ 7 days.

SUMMARY:
To date, there are highly effective lipid-lowering drugs, the combination of which makes it possible to achieve the target level of LDL-C in most patients with familial hypercholesterolemia (FH). However, the effectiveness of treatment of FH patients strongly depends on adherence to lipid-lowering therapy and to the healthy lifestyle, as well as the detection of the disease and the therapy prescription as early as possible, better in childhood. The aim of the study is to assess the impact of genetic testing and motivational counseling on the effectiveness of treatment and cascade screening in patients with FH.

DETAILED DESCRIPTION:
There are several tasks of the study:

1. To assess the effect of knowledge of patients with FH about the result of their FH genetic testing on the adherence to a healthy lifestyle and hypolipidemic therapy.
2. To assess the impact of knowledge of patients with FH about the result of their FH genetic testing on the effectiveness of cascade screening.
3. To assess the influence of motivational counseling of patients with FH on the adherence to a healthy lifestyle and hypolipidemic therapy.
4. To assess the impact of motivational counseling of patients with FH on the effectiveness of cascade screening.

ELIGIBILITY:
Inclusion Criteria:

* Probable or definite diagnosis of FH according to the Dutch criteria (6 points or more);
* Signed informed consent;

Exclusion Criteria:

* Pregnancy or lactation at the time of enrollment
* Established active severe infectious disease or severe hematologic, metabolic, gastrointestinal or endocrine dysfunctions (for example, uncontrolled thyroid dysfunction or uncontrolled diabetes mellitus) in the opinion of the investigator
* Active liver disease
* Estimated GFR≤ 30 ml / min / 1.73m2
* Any other conditions at Visit 1 that, according to the investigator's opinion, render the patient ineligible for inclusion in the study, may interfere with the patient's participation in the study or patient's completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in the proportion of people who have reached the target level of LDL-Cholesterol | 3 months
  Change in the proportion of people who have reached the target level of LDL-Cholesterol (target values of LDL-C according to the ESC Dislipidaemia Guidelines 2019)
Change in the number of relatives who underwent cascade screening | 3 months
  Change in the number of relatives who underwent cascade screening (% of relatives out of all available relatives. Available relatives are those who are alive and live in the region of where the study is conducted (Moscow and Moscow region)
Change in the proportion of people adhering to drug therapy | 3 months
  Change in the proportion of people adhering to drug therapy according to the questionnaire MARS-5
Change in the proportion of people adhering to the recommended physical activity | 3 months
  Change in the proportion of people adhering to the recommended physical activity (according to the Global Physical Activity Questionnaire (GPAQ))
Change in the proportion of individuals adhering to the recommended dietary recommendations | 3 months
  Change in the proportion of individuals adhering to the recommended dietary recommendations (according to 24-hour Dietary Recall and Food Frequency Questionnaires)

SECONDARY OUTCOMES:
Change in the proportion of people who have reached the target level of LDL-Cholesterol | 15 months
  Change in the proportion of people who have reached the target level of LDL-Cholesterol (target values of LDL-C according to the ESC Dislipidaemia Guidelines 2019)
Change in the number of relatives who underwent cascade screening | 15 months
  Change in the number of relatives who underwent cascade screening (% of relatives out of all available relatives. Available relatives are those who are alive and live in the region of where the study is conducted (Moscow and Moscow region)
Change in the proportion of people adhering to drug therapy | 15 months
  Change in the proportion of people adhering to drug therapy according to the questionnaire MARS-5
Change in the proportion of people adhering to the recommended physical activity | 15 months
  Change in the proportion of people adhering to the recommended physical activity (according to the Global Physical Activity Questionnaire (GPAQ))
Change in the proportion of individuals adhering to the recommended dietary recommendations | 15 months
  Change in the proportion of individuals adhering to the recommended dietary recommendations (according to 24-hour Dietary Recall and Food Frequency Questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Meshkov, MD, PhD, Principal Investigator — National Medical Research Centre for Therapy and Preventive Medicine, Ministry of Health of Russia; Alexandra Ershova, MD, PhD, Study Director — National Medical Research Centre for Therapy and Preventive Medicine, Ministry of Health of Russia
Locations (1):
- National Medical Research Centre for Therapy and Preventive Medicine of the Ministry of Health of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blokhina AV, Ershova AI, Kopylova OV, Limonova AS, Karamnova NS, Shvabskaya OB, Kiseleva AV, Derbeneva SA, Meshkov AN, Drapkina OM. [Actual nutrition in adults with familial hypercholesterolemia]. Vopr Pitan. 2023;92(4):49-58. doi: 10.33029/0042-8833-2023-92-4-49-58. Epub 2023 Jun 30. Russian. PMID 37801454